CLINICAL TRIAL: NCT06097988
Title: A Prospective, Multicenter Clinical Investigation Evaluating the Safety of ABIO3419 in Treating Knee Osteoarthritis: Pilot Study
Brief Title: Study on Knee Osteoarthritis
Acronym: PILHAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2301
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABIO3419 (Experimental): Patients will be included consecutively to receive ABIO3419 by intra-articular injection
  Interventions: Device: ABIO3419

INTERVENTIONS:
Device: ABIO3419 — Intra-articular injection

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative joint disease characterized macroscopically by progressive damage of articular cartilage, joint space narrowing, subchondral bone remodelling, joint marginal osteophyte formation and synovitis. It is also characterized by a decrease of the concentration and molecular weight of the hyaluronic acid in the synovial fluid which ultimately leads to poor viscoelastic properties of synovial fluid and induction of proinflammatory pathways.

The intra-articular injection of viscosupplementation gel (mainly exogenous hyaluronic acid) represents one of the most used therapeutic strategies to treat osteoarthritis symptoms.

Several studies on knee Osteoarthritis, have shown that one or more weekly injection of viscosupplementation gel significantly relieves articular pain and ameliorates mobility and joint function for at least 6 months and more. Repeated courses of intra-articular injections are an effective and safe treatment for knee osteoarthritis symptoms.

Based on studies conducted on intra-articular viscosupplementation gels, the most common side effects expected are local transient and short-lived adverse events such as pain, swelling and arthralgia in the site of administration, which are fully reversible in the days following the injection. Furthermore, such local effects may occur in a minority of cases and are usually treated conservatively with ice, non-steroidal anti-inflammatory drugs, and relative rest.

DETAILED DESCRIPTION:
The study is a pilot, prospective, multicenter, clinical trial that aims to evaluate the safety and efficacy of ABIO3419 for the treatment of knee osteoarthrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily given informed consent to investigation participation in writing encompassing consent to data recording and verification procedures.
2. Male and female subjects, aged 35 to 85 years (inclusive).
3. Subjects affected by knee osteoarthritis, as defined by American College of Rheumatology (ACR) clinical and radiographic criteria for osteoarthritis of the knee, and meeting the following conditions:

   1. Kellgren-Lawrence Grade 2 to 3 severity osteoarthritis of the knee confirmed by an extension face X-rays shot, supported by flexion face X-rays shot (optional) obtained within 6 months from the screening visit.
   2. Subjects suffering from osteoarthritis symptoms of the target knee for at least 6 months prior to the screening visit.
4. Pain during walking on flat ground in the target knee of at least 40 mm and maximum 80 mm on a 0-100 mm Visual Analogic Scale at the baseline visit (Visit 2).
5. Women of childbearing potential must have a negative urine pregnancy test prior to each injection.
6. Subject who is able to comply with the study requirements, at the Investigator's appreciation.
7. Subject being affiliated to a health social security system

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Subject with bilateral osteoarthritis of the knees is excluded if one of the following point is present on the non-targeted knee has:

   * a visual analog scale score greater than 30mm (> 30mm),
   * a Kellgren-Lawrence score is greater than 2 (>2)
   * a dedicated antalgic consumption.
3. Subject suffering from a severe or progressive disease or any other pathology which, according to the investigator, may interfere with evaluation of the results of the study: diabetes, autoimmune pathology, cardiac pathologies, hepatic deficiency, epilepsy, porphyria, rheumatoid arthritis or other systemic inflammatory process.
4. Subject who has a known history of severe multiple allergies, angioedema or anaphylactic shock according to the investigator opinion.
5. Subject with a known allergy or hypersensitivity to Hyaluronic Acid or bovine collagen.
6. Subject with a past history of severe streptococcal disease or an active streptococcus infection according to the investigator opinion.
7. Subject with a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
8. Subject having received chemotherapy agents, immunosuppressive medications within the past 3 months.
9. Subject with bleeding disorders or subject received medication (anti-platelet agents and anticoagulant) that will likely increase the risk of bleeding within the past 24 hours before injections.
10. Subjects having received:

    1. Intra-articular knee corticosteroids within 60 days prior to the baseline visit.
    2. Chondroitinsulphate, glucosamine sulphate, diacereine, bisphosphonates or matrix metalloproteinase inhibitors within 30 days prior to the baseline visit.
    3. Viscosupplementation of the target knee within 6 months prior to the baseline visit.
    4. Any kind of antalgic and Non-steroidal anti-inflammatory drugs in the 24 hours prior to the baseline visit (V2) and before each visit.
11. Subjects with a Kellgren-Lawrence grade 4 femora-patellar osteoarthritis or subjects with a femora-patellar osteoarthritis Kellgren-Lawrence grade higher than the femora-tibial one.
12. Subjects with coxarthrosis.
13. Subjects having had any previous surgery in the target knee within 6 months prior to the screening visit, or any planned surgery in the target knee throughout the duration of the investigation.
14. Subjects who have had arthroplasty at the target knee at any time.
15. Subjects having had diagnostic or surgical knee arthroscopy, or knee lavage in the target knee in the 6 months prior to the screening visit.
16. Subjects that are candidate for knee replacement within next 6 months.
17. Subjects with body mass index > 35 kg/m2.
18. Subjects with large intra-articular effusion of the target knee, venous or lymphatic stasis, inflammatory flare-up with various symptoms, local inflammation.
19. Subjects with history of septic osteoarthritis of any joint
20. Subjects with significant pain outside the target knee, including significant hip or back pain and with fibromyalgia.
21. Subjects with clinically significant valgus/varus deformities, ligamentous laxity, or meniscal instability as assessed by the Investigator.
22. Subjects with other musculoskeletal condition affecting the target knee that would impair assessment of the effectiveness in the target knee (e.g. Paget's disease of bone).
23. Subjects with a current malignancy or having treatment for a malignancy, except non-melanoma skin cancer.
24. Subjects with drug or alcohol abuse
25. Subject who is deprived of their freedom by administrative or legal decision.
26. Subject living in a social or sanitary establishment.
27. Subject being in an exclusion period for a previous study or with a current or recent (<3 months) participation in another investigational study involving a drug or combined device with drug.
28. Other condition preventing the subject to participate the study in the Investigator's opinion: subject deemed unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment results.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse device effects related to ABIO34199 treatment [tolerability] at 3 months | Month 3 after the last injection
  Assessment by the investigators of the occurrence of adverse device effects related to ABIO3419 from the first injection up to the 3-month follow-up

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | Immediately after first injection, before and immediately after the injections at 1 week and 2 weeks, then at 2 weeks, 1 month, 3 months and 6 months after the last injection
  Collection of Adverse Event assessed and recorded by investigators.
Evaluation of the pain of the treated knee when walking on a flat ground. | Baseline (before initial injection), 1 week and 2 weeks after the first injection (before 2nd and 3rd injections) then 2 weeks, 1 month and 3 months after the last injection.
  Assessment by the patient itself of the pain compared to baseline (before initial injection) using a 0-100mm Visual Analogue Scale (0 corresponds to no pain and 100 corresponds to the highest pain that can be felt).
Device related complication rates | Immediately after first injection, before and immediately after the injections at 1 week and 2 weeks, then at 2 weeks, 1 month, 3 months and 6 months after the last injection
  Assessment of the proportion of patient with at least one adverse device effect related to ABIO3419 at each time visits
General health status of the treated knee | Baseline (before initial injection), 1 week and 2 weeks after the first injection (before 2nd and 3rd injections) then 2 weeks, 1 month and 3 months after the last injection.
  Assessment by the patient itself of the target-knee functional status using the Knee injury and Osteoarthritis Outcome Score (KOOS).
  The KOOS holds 42 items in 5 separately scored subscales: Pain (nine items); Symptoms (seven items); Function in daily living (17 items); Sport and Recreation Function (five items); Quality of Life (four items).
  A 5-grade Likert scale is used for all items scored from 0 (No Problems) to 4 (Extreme Problems).
  Each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Concomitant analgesic consumption | 1 week before the first injection, 1 week and 2 weeks after the first injection then 2 weeks, 1 month and 3 months after the last injection.
  Assessment by the patient of the average weekly consumption (number and dosage) of paracetamol and pain killer drugs using a daily diary.
Implant card readability | Day 0 (after first injection)
  Assessment of the patient of the reading and understanding of the ABIO3419 implant card using a questionnaire on which the text present on the implant card must be identified and reported on the questionnaire.
Investigator Global satisfaction | Week 2 after first injection
  Assessement by the investigator of the handling of the ABIO3419 device with a Usability questionnaire after the third injection with four response possibilities for each item: Very satisfied / Satisfied / Neutral / Not satisfied.
Investigator Global satisfaction | Month 6
  Assessement by the investigator of the overall satisfaction with a satisfaction questionnaire at 6 months with four response possibilities for each item: Very satisfied / Satisfied / Neutral / Not satisfied.
Patient Global satisfaction | month 6
  Assessement by the patient of the overall satisfaction with a satisfaction questionnaire at 6 months with four response possibilities for each item: Very satisfied / Satisfied / Neutral / Not satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kristaps KNOHENFELDS, Principal Investigator — Veselibas Centrs ZIN; Kalvis KRASTINS, Principal Investigator — Private Office Centrs
Locations (2):
- Latvia (2):
  - Knohenfelds, Riga, Rīga
  - KRASTINS, Riga, Rīga